CLINICAL TRIAL: NCT04015401
Title: Neuropathic Pain in Jamaicans With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: The University of The West Indies (Other)
Collaborators: Avicanna Inc (Industry)
Responsible Party: Principal Investigator, Monika Parshad-Asnani, Senior Lecturer, The University of The West Indies
Other Study IDs: NP001
Record Dates: First submitted 2019-07-04; First posted 2019-07-11 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Sickle Cell Disease; Neuropathic Pain
Keywords: Quantitative sensory testing; Jamaica
MeSH Terms: conditions — Anemia, Sickle Cell; Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pain is the most common component of the morbidity seen in sickle cell disease (SCD), and may be acute or chronic. It is most commonly acute and a result of the hallmark vaso-occlusive episodes of the disease. Many patients however suffer from chronic pain - defined as pain lasting over three months- with neuropathic pain being a component of chronic pain. Neuropathic pain significantly contributes to the chronicity and morbidity of pain in SCD patients, and is an inadequately managed complication. There is a paucity of literature covering this area, and it has never been examined in the Jamaican population. The main objective of this study is to determine the epidemiology of pain among Jamaicans with SCD, and determine the prevalence of chronic and neuropathic pain among these patients. A second objective is to validate, using gold-standard measures, screening tools to determine neuropathic pain among the study population. This cross-sectional study will investigate the prevalence of neuropathic pain and complications in a sample of persons with SCD in Jamaica aged 14 years and older, with a validation sub-study to be conducted on a random 20 percent of the sample. With improved diagnosis of neuropathic pain, clinicians may potentially improve the management of pain in SCD, as clinicians should be able to direct our treatment toward medications and non-pharmacological methods of pain relief that are more specific for neuropathic pain. All data will be de-identified and maintained in a secure database, with access limited to key personnel. There is very minimal risk to participants.

DETAILED DESCRIPTION:
All study participants will complete all the questionnaires provided, specifically the Adult Sickle Cell Quality of Life Measurement Information (ASCQ-Me), Leeds Assessment of Neuropathic Symptoms and Signs (LANSS), PainDETECT and Douleur Neuropathique 4 (DN4). All study participants will also have qualitative sensory testing and laboratory investigations done. Nerve conduction studies will only be done on a randomly selected 20 percent sub-study sample.

Laboratory investigations include sample of blood (~ 10 mls) will also be collected for the participants and analysed for Haemoglobin (steady state), white blood cells, and lactate dehydrogenase, percent reticulocytes. These are common markers of disease severity in SCD. Disease severity is one of the variables which will be used in the epidemiological description of the study population as well as in the statistical analysis of the data.

The Q-Sense will be used to conduct quantitative sensory tests. This allows specific degrees of heat/cold stimulation to assess sensation and pain thresholds to be applied and patients indicate at which degree they detect the stimuli and furthermore when it becomes painful, at each site. The results are then compared to known controls. Hypersensitivity and allodynia to thermal stimuli is considered diagnostic for neuropathic pain. The tests are considered safe in sickle cell patients and when tested have not resulted in any crisis. Patients may experience mild pain after the test, and therefore will be asked to take their regular analgesics immediately following the test.

Nerve conduction studies (NCS): A subset of participants identified with chronic or presumed neuropathic pain will, in addition to QST, receive a standard neurophysiological evaluation by nerve conduction studies to determine the presence/absence of a large fibre neuropathy, whether a focal mononeuropathy or diffuse polyneuropathy. Polyneuropathies will be characterized by process as either axonal or demyelinating, and by pattern as sensory, motor or sensorimotor, with comparisons to findings on QST.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 14 and older, of any sex and genotype
* Informed consent/parental consent with child assent available
* In well state at time of study

Exclusion Criteria:

* Prior cerebrovascular accidents
* Acute illness at time of recruitment
* Current Pregnancy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Using the Sickle Cell Unit (SCU) of the University of the West Indies patient management system, a computer generated random selection of the sample will be carried out from a sampling frame of all patients aged 14 years and older who are coded as 'alive' upon last visit, and who have had at least one visit to the SCU in the last 2 years. The recruitment of participants to satisfy the sample size of 528 participants will be stratified according to five age-sex categories i.e. male and female 14 - 24; 25 - 34; 35 - 44; 45 - 54; 55 + years old. Selected participants will be recruited by phone to attend a clinic appointment where informed consent will be ascertained.
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of neuropathic pain among Jamaicans with Sickle cell disease (SCD) | 1 year
  Determine among a clinic population of persons with SCD the prevalence of chronic and neuropathic pain

SECONDARY OUTCOMES:
Effect of age on neuropathic pain | 1 year
  Is age ( in years) correlated with the presence of neuropathic pain in persons with SCD
Effect of sex on neuropathic pain | 1 year
  Is sex (male or female) correlated with the presence of neuropathic pain in persons with SCD

OTHER OUTCOMES:
Validation of common screening tool, PainDetect, in detection of neuropathic pain in persons with sickle cell disease | 1 year
  Determine limits of agreement of detecting the presence of neuropathic pain using common screening tools with the gold standard measurement using quantitative sensory testing

CONTACTS AND LOCATIONS:
Overall Officials: Monika Asnani, DM PhD, Principal Investigator — Caribbean Institute for Health Research; Zachary Ramsay, MBBS, Study Director — Caribbean Institute for Health Research
Locations (1):
- Caribbean Institute for Health Research, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: No